CLINICAL TRIAL: NCT07305584
Title: Regional Anesthesia for Elderly Patients Undergoing Distal Upper Limb Surgeries: A Randomized Comparative Study of Subcoracoid Tunnel Block Versus Costoclavicular Block
Brief Title: Comparative Study of Subcoracoid Tunnel Block Versus Costoclavicular Block
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Marwa Mohamed Medhat, assistant professor of anesthesia and surgical intensive care(Principal Investigator), Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZU-IRB#1885/7-Nov-2025
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Distal Upper Limb Surgeries
Keywords: distal Upper Limb Surgeries Subcoracoid Tunnel Block Costoclavicular Block

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (S) (Active Comparator): The patient will receive subcoracoid tunnel block
  Interventions: Other: subcoracoid tunnel block
- Group (C) (Active Comparator): The patient will receive costoclavicular block
  Interventions: Other: Costoclavicular block

INTERVENTIONS:
Other: subcoracoid tunnel block — The probe will be placed with its proximal end towards the mid-clavicular point and distal end with a marker towards the apex of the axilla. A medial tilt of the probe will demonstrate the posterior and medial cords, while a slight lateral tilt of the probe will demonstrate the lateral cord. The needle entry point at the distal end of the probe will be marked. By using the in-plane technique, the needle will be advanced from a caudal to cephalad direction. The probe will be tilted medially, and the needle will be advanced to position its tip above the posterior or medial cord. The probe will be tilted laterally. The needle tip will be repositioned above the lateral cord, and the LA will be injected
  Arms: Group (S)
Other: Costoclavicular block — . The key anatomical structures will be identified under ultrasound: the pectoralis major muscle, subclavius muscle, and three brachial plexus cords (lateral, medial, and posterior) clustered tightly lateral to the axillary artery, along with the axillary artery and vein. The needle will be inserted by the in-plane technique from lateral to medial. The needle tip will be advanced through subcutaneous tissue and subclavius, aiming to land in the costoclavicular fascial plane between the cords, ideally between the lateral and posterior cords and superficial to the medial cord, without traversing neural structure by multipoint strategy, and local anesthesia will be injected.
  Arms: Group (C)

SUMMARY:
The purpose of this study is to compare the analgesic outcomes (time to first analgesic request, total amount of analgesic consumption, and pain scores) following the ultrasound-guided subcoracoid tunnel block or costoclavicular block for elderly patients undergoing distal upper limb surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Patients acceptance to share in the study.
* Patients with ASA physical status I-II.
* Patients with a body mass index (BMI): of 18.5-30 kg/m2.
* Patients undergoing distal upper limb surgeries not more than 2 hours.

Exclusion Criteria:

* Patients with a history of allergic reactions or contraindications to local anesthetics.
* Patients with significant comorbidities (e.g., severe cardiovascular, neurological, or musculoskeletal disorders).
* Patients with respiratory insufficiency.
* Patients with coagulation disorders or taking drugs affecting surgical hemostasis.
* Patients with pre-existing neurological deficits

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
the onset time of sensory block | 5 minutes after the block
  the time interval between the end of total local anesthetic administration and complete sensory block

SECONDARY OUTCOMES:
block performance time | time of performance of the block
3. Time of first rescue analgesia(naluphine) | 24 hours postoperative
Pain intensity | basal, one, 2, 4, 8, 12, 18, 24, and 24 hours postoperative
  10-point NRS [(0 = no pain, 10 = worst imaginable pain), 1-3: Mild pain (nagging, annoying, slightly interfering with activities of daily living (ADLs), 4 - 6: Moderate pain (significantly interfering with ADLs, 7 - 10: Severe pain (disabling, unable to perform ADLs)]
patient's satisfaction | 24 hours postoperative
  The patients will be asked to rate the overall degree of satisfaction of the analgesia by using a 5-points likert-like verbal scale (1 = very dissatisfied analgesia, 2 = dissatisfied analgesia, and 3 = neutral, 4=satisfied analgesia, and 5=very satisfied analgesia)
Incidence of block complications | first 24 hours postoperative
  hematoma formation or paresthesia or local anesthetic systemic toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Howida A Kamal, MD, Study Director — faculty of medicine,zagazig university Egypt
Locations (1):
- faculty of medicine,zagazig university Egypt, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kaya S, Sahap M, Demirtas K. Comparison of costoclavicular and lateral sagittal infraclavicular approaches in ultrasound-guided brachial plexus block. Agri. 2025 Jan;37(1):32-41. doi: 10.14744/agri.2024.34022. PMID 39835953